CLINICAL TRIAL: NCT05715411
Title: Assessment of Light Therapy in Insomnia Disorder
Acronym: InsomLum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7680
Record Dates: First submitted 2023-01-04; First posted 2023-02-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Other: Placebo with light therapy glasses
- Light therapy (Experimental)
  Interventions: Other: light therapy with light therapy glasses

INTERVENTIONS:
Other: Placebo with light therapy glasses — Placebo
  Arms: Control
Other: light therapy with light therapy glasses — light therapy
  Arms: Light therapy

SUMMARY:
Sleep disorders represent a major public health issue and the leader in these disorders is insomnia with 10 to 15% of subjects in the general population reporting symptoms of insomnia with a daytime impact. In addition to being very common, insomnia leads to an increase in morbidity and mortality and weighs on healthcare systems worldwide. Despite this public health context, insomnia is underdiagnosed and rarely treated. Hypnotics have proven efficacy but with a risk of dependence and pharmacotolerance which appears within a few weeks. Cognitive behavioral therapy (CBT) has a good level of evidence and is now a benchmark treatment for the management of insomnia. Unfortunately, not all patients adhere to or respond to these procedures, which cannot be implemented for many of them either. There is therefore a need to identify other alternative therapeutic strategies, and we believe that exposure to light is a promising treatment.

In this perspective, it seems interesting to assess the effect of the propensity to fall asleep with an exposure to light therapy in patients suffering from insomnia.

In order to be in optimal ecological conditions, we want to use a portable light therapy device which allows easy, acceptable and ambulatory exposure.

If the lighttherapy is confirmed in insomnia under ecological conditions, this would make it possible to propose a new non-drug treatment, easy to access and on a large scale

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 30 to 60 years
* Insomnia disorders (ICSD-3) with sleep latency >30min - 3 times a week
* Patient able to understand the objectives and risks associated with the research and to give informed dated and signed consent
* Patient affiliated to a social health insurance scheme
* For women of childbearing age, effective contraceptive measure for the duration of the research (hormonal contraception, IUD).

Exclusion Criteria:

* - Shift work in the year preceding inclusion
* Trans meridian travel (> 2 time zones) in the month preceding inclusion
* Patient in exclusion period determined by a previous or ongoing study
* Impossibility of giving the patient informed information (emergency patient, difficulty understanding the patient)
* Patient under judicial protection
* Patient under guardianship or curatorship
* For a woman of childbearing age: ongoing pregnancy or breastfeeding
* Drug treatment which can disturb sleep or the measurement of DLMO: corticosteroids by general route, beta-blockers in the evening, exogenous melatonin.
* Phase delay syndrome defined according to the criteria of the international classification of ICSD-3
* Restless legs syndrome with IRLS score> 20
* Other psychiatric disorders or addictive disorder (screening with the MINI structured interview)
* Other medical conditions not stabilized (detected by clinical interview), only the diseases appearing in the following list will constitute a criterion of non-inclusion:

  * Chronic allergies
  * Neurological disorders
  * cardiovascular, respiratory, gastrointestinal, hematopoietic, visual diseases
  * diseases of the immune system
  * kidney and urinary tract diseases
  * endocrine and metabolic diseases
  * infectious diseases
  * epilepsy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change Sleep latency | At day 0 and Day 44
  Actimetry is used to compare the sleep latency

SECONDARY OUTCOMES:
Change Daytime sleepiness | At day 0 and Day 90
  Epworth Scale is used to compare the sleepiness in baseline to completion of the procedure and three month after intervention
Change Daytime sleepiness | At day 0 and Day 90
  Karolinska Sleepiness Scale is used to compare the sleepiness in baseline to completion of the procedure and three month after intervention
Change Circadian rythms | At day 0 and Day 90
  Circadian markers melatonin is measured in baseline, completion of the procedure and three month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrice BOURGIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No